CLINICAL TRIAL: NCT05545800
Title: Efficacy and Safety Of Different Hypoglycemic Regimens Compared With Premixed Insulin In Patients With Type 2 Diabetes Receiving Short-term Intensive Insulin Therapy
Brief Title: Efficacy and Safety Of Different Regimens In Patients With Type 2 Diabetes Receiving Intensive Insulin Therapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202206361
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — IDegLira

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- metformin+empagliflozin+insulin glargine (Experimental): metformin+empagliflozin+insulin glargine
  Interventions: Drug: metformin+empagliflozin+insulin glargine
- IDegLira (Experimental): IDegLira
  Interventions: Drug: IDegLira
- premixed insulin analogues (Active Comparator): premixed insulin analogues
  Interventions: Drug: premixed insulin analogues

INTERVENTIONS:
Drug: metformin+empagliflozin+insulin glargine — Randomization was performed with the use of a computer-generated system provided by the sponsor. The dose of metformin will be initiated at 0.5 grams three times a day (the maximum dose is 2g/day); the dose of empagliflozin will be 10 milligrams once a day; insulin glargine will be received once daily at bedtime and the dose will be initiated at the 50% of 0.4-0.5 units/kg/day. All groups received counseling on lifestyle modification.
  Arms: metformin+empagliflozin+insulin glargine
Drug: IDegLira — Randomization was performed with the use of a computer-generated system provided by the sponsor. Eligible patients will be initiated on 16 units (16 units degludec/0.58 mg liraglutide) and titrated twice weekly. The maximum dose of IDegLira was 50 units (50 units degludec/1.8 mg liraglutide). All groups received counseling on lifestyle modification.
  Arms: IDegLira
Drug: premixed insulin analogues — Randomization was performed with the use of a computer-generated system provided by the sponsor. Eligible patients will received twice a day. The total daily insulin dose will be initiated at 0.4-0.5 units/kg/day and adjusted according to the plasma glucose. All groups received counseling on lifestyle modification.
  Arms: premixed insulin analogues

SUMMARY:
The purpose of this studay is to compare the efficacy of different hypoglycemic regimens versus twice-daily premixed insulin in type 2 diabetes mellitus (T2DM) patients after short-term ntensive Insulin Therapy by using continuous glucose monitoring.

DETAILED DESCRIPTION:
This randomized, positive-controlled, open-label, parallel-group study will enroll approximately 78 male and female patients aged 18-70 years with poorly-controlled T2DM (HbA1c >9% or FBS>11.1mmol/L) after short-term intensive insulin therapy. Eligible patients will then be randomized in a 1:1:1 ratio to insulin glargine plus OADs or twice-daily premixed insulin or Insulin Degludec & Liraglutide for 3 months with metformin maintained throughout the study in both treatment groups. All the patients will wear CGM during short-term intensive insulin therapy and after treatment for 7 days. The primary endpoint is plasma glucose change from baseline to month 3. Secondary endpoints include assessment of fasting plasma glucose, total daily insulin dose, hypoglycemia incidence, body weight change, adverse events, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-70 years with poorly-controlled T2DM (World Health Organization diagnostic criteria)
* BMI 21~32Kg/m2
* duration of T2DM more than 1 year
* FPG≥11.1mmol/L or HbA1c ≥9% for three months
* fasting C-peptide >1 ng/mL

Exclusion Criteria:

* acute diabetic complications (diabetic ketoacidosis, lactic acidosis, hyperosmolar nonketotic diabetic coma) within the past 1 month;
* impaired renal function,defined as (but not limited to) serum creatinine levels ≥1.5 mg/dL for males and ≥1.4 mg/dL for females, or the presence of macroproteinuria (> 2 g/day)
* pregnancy
* inability to perform self-monitoring of BG (SMBG)
* acute disease or surgery in the past 3months or preparation for the surgey

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Mean Change From Baseline in HbA1c | Month 0 to 3
  mean change from baseline in HbA1c after 3-months of treatment.
Percentage of patients achieving HbA1c <7% | Month 0 to 3
  Percentage of patients achieving HbA1c <7% after 3-months of treatment.
Amplitude of glycemic excursions | Month 0 to 3
  Amplitude of glycemic excursions from month 0 to 3

SECONDARY OUTCOMES:
Percentage of hypoglycemia incidence | Month 0 to 3
  Percentage of hypoglycemia incidence from month 0 to 3
Percentage of adverse events | Month 0 to 3
  Percentage of adverse events from month 0 to 3

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wu, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China